CLINICAL TRIAL: NCT01474616
Title: Mobility of Vulnerable Elders (MOVE): Translating Knowledge to Health Care Aides in Long-term Care Facilities
Acronym: MOVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CapitalCare Continuing Care (Unknown); Extendicare (Unknown); Good Samaritan Society (Unknown); Shepherd's Care Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DPA 108891
Record Dates: First submitted 2011-11-10; First posted 2011-11-18 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2013-07

CONDITIONS: Mobility Limitation
Keywords: Aging; Health Services; Knowledge Translation; Long-Term Care Facilities; Mobility; Psychosocial And Health Behaviours
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sit-to-Stand Activity (Other)
  Interventions: Other: Sit-to-Stand Activity

INTERVENTIONS:
Other: Sit-to-Stand Activity — Health care aides will be expected to prompt residents to repeatedly stand up and sit down on four occasions throughout the day (twice on each of the day and evening shifts). The number of repetitions on each occasion will vary according to residents' ability and fatigue. The sit-to-stand activity is to be integrated into usual care routines such as when entering the dining room at mealtimes, while toileting, and on other occasions of regular activity. The timing and location will be at the discretion of the health care aide.

SUMMARY:
Almost 90 percent of residents living in long-term care facilities have some type of mobility limitation, which worsens quickly once they move into a long-term care facility. This means that they cannot easily walk or move around in their day-to-day lives and this can have serious consequences for their general health and well-being. Researchers have shown that exercise can help the mobility of even the oldest of adults but elderly residents in long-term care facilities still commonly sit or lie in bed for long periods of time, in many cases for most of their waking hours. The purpose of this research is to study the effect of a simple physical activity on the mobility and quality of life of residents in long-term care facilities. Researchers will introduce a sit-to-stand activity to health care aides which will become part of their daily routine with residents. The basic sit-to-stand movement is already a part of the daily activities that health care aides do with residents. Specifically, health care aides will ask residents to repeat the sit-to-stand activity at mealtimes, when using the toilet, and on other occasions of daily activity. An important part of this research is to find out how well the activity preserves the ability of residents to stay mobile and also to examine how this will improve their quality of life in the home. The MOVE study will demonstrate whether it is possible to delay the loss of mobility in long-term care residents by incorporating the sit-to-stand activity into the regular practice of health care aides.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of Alzheimer disease, vascular dementia, or mixed dementia
* are able to transfer independently or with the assistance of one person

Exclusion Criteria:

* have a diagnosis of fronto-temporal or Lewy-body dementia
* require the assistance of more than one person to transfer, or a transfer lift

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Mobility at 3 and 6 months | Baseline, 3-Months, 6-Months
  The sit-to-stand action is a functional activity that has been incorporated into a number of mobility measures. We have chosen to measure mobility using the number of sit-to-stands in 30 seconds because in the frail nursing home population many residents have difficulty transferring (e.g.standing up from a chair). In our pilot study we found many residents were unable to complete more than two or three sit-to-stands. Residents will be instructed to stand up and sit down as many times as possible until they are asked to stop after 30 seconds (Jones, Rikli, & Beam, 1999).

SECONDARY OUTCOMES:
Change from Baseline in Function at 3 and 6 months | Baseline, 3-Months, 6-Months
  The Functional Independence Measure (FIM) is an 18-item performance-based instrument which assesses the amount of assistance required to complete basic activities of daily living using a 7-point scale graded from 1 (dependent) to 7 (independent) (Jones & Feeny, 2006).
Change from Baseline in Health Related Quality of Life at 3 and 6 months | Baseline, 3-Months, 6-Months
  The Health Utilities Index Mark 2 and 3 (HUI2/3) is a generic health related quality of life questionnaire based on two generic multi-attribute preference-based systems: the HUI2 and the HUI3. The HUI2 assesses capacity on six dimensions (or attributes) of health status: sensation (vision, hearing, and speech), mobility, emotion, cognition, self-care, and pain. The HUI3 consists of eight attributes: vision; hearing; speech; ambulation; dexterity; emotion; cognition; and, pain (Furlong, et al., 2011).
Change from Baseline in Dementia Specific Quality of Life at 3 and 6 Months | Baseline, 3-Months, 6-Months
  The Quality of Life-Alzheimer's Disease (QofL-AD) was developed to capture the domains considered important to quality of life in Lawton's broad conceptual framework: the interpersonal; environmental; functional; physical; and, psychological domains. The 13 items including physical health, energy, mood, living situation, memory, family, marriage, friends, self as a whole, ability to do chores around the house, fun, money, life as a whole scored on a 4-point Likert scale ranging from 1 (poor) to 4 (excellent) (Lawton, 1983; 1991).

CONTACTS AND LOCATIONS:
Overall Officials: Susan Slaughter, RN, PhD, Principal Investigator — University of Alberta
Locations (4):
- Canada (4):
  - CapitalCare Continuing Care, Edmonton, Alberta
  - Good Samaritan Society, Edmonton, Alberta
  - Extendicare, Edmonton, Alberta
  - Shepherd's Care Foundation, Edmonton, Alberta

REFERENCES:
- [Result] Slaughter SE, Wagg AS, Jones CA, Schopflocher D, Ickert C, Bampton E, Jantz A, Milke D, Schalm C, Lycar C, Estabrooks CA. Mobility of Vulnerable Elders study: effect of the sit-to-stand activity on mobility, function, and quality of life. J Am Med Dir Assoc. 2015 Feb;16(2):138-43. doi: 10.1016/j.jamda.2014.07.020. Epub 2014 Sep 27. PMID 25271194
- [Derived] Slaughter SE, Estabrooks CA, Jones CA, Wagg AS. Mobility of Vulnerable Elders (MOVE): study protocol to evaluate the implementation and outcomes of a mobility intervention in long-term care facilities. BMC Geriatr. 2011 Dec 16;11:84. doi: 10.1186/1471-2318-11-84. PMID 22176583